CLINICAL TRIAL: NCT00122902
Title: Spirituality and Will to Live in Patients With HIV/AIDS
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: R01AT001147-01 (NIH)
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Spirituality
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study is assessing the extent of spirituality in patients with HIV/AIDS and will determine the relationship between spirituality, health status, and the will to live.

DETAILED DESCRIPTION:
Approximately 1,000,000 Americans have HIV/AIDS. Although advances in treatment have made HIV/AIDS a relatively manageable chronic disease, the disease can cause significant morbidity and mortality. Surprisingly, research has found that some HIV/AIDS patients feel that their life is better than it was before they had HIV/AIDS. Many of these patients show a strong will to live and often express a preference for longevity over quality of life. Patients who prefer longevity often ascribe their feeling to spiritual growth, or finding a meaning to life. This study is examining the spiritual beliefs of HIV/AIDS patients and will determine the relationship between spirituality, health status, and the will to live.

The study consists of interviews with HIV/AIDS patients from Cincinnati and Washington, D.C. who have been interviewed twice over 12 to 18 months. During the interviews, participants completed self-report scales to assess their quality of life, life satisfaction, concerns about medication, trust in their health care providers, depressive symptoms, self-esteem, optimism, and various clinical and demographic variables. Participants were also asked about their spiritual well-being; spiritual beliefs; spiritual, religious, and social support; and overall functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV or AIDS

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2002-02; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Joel Tsevat, MD, MPH, Principal Investigator — Division of General Internal Medicine, University of Cincinnati Medical Center
Locations (1):
- Division of General Internal Medicine, University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Luckhaupt SE, Yi MS, Mueller CV, Mrus JM, Peterman AH, Puchalski CM, Tsevat J. Beliefs of primary care residents regarding spirituality and religion in clinical encounters with patients: a study at a midwestern U.S. teaching institution. Acad Med. 2005 Jun;80(6):560-70. doi: 10.1097/00001888-200506000-00011. PMID 15917361
- [Background] Yi MS, Luckhaupt S, Mrus JM, Tsevat J. Do medical house officers value the health of veterans differently from the health of non-veterans? Health Qual Life Outcomes. 2004 Apr 7;2:19. doi: 10.1186/1477-7525-2-19. PMID 15070409
- [Result] Mrus JM, Yi MS, Freedberg KA, Wu AW, Zackin R, Gorski H, Tsevat J. Utilities derived from visual analog scale scores in patients with HIV/AIDS. Med Decis Making. 2003 Sep-Oct;23(5):414-21. doi: 10.1177/0272989X03256884. PMID 14570299
- [Result] Mrus JM, Sherman KE, Leonard AC, Sherman SN, Mandell KL, Tsevat J. Health values of patients coinfected with HIV/hepatitis C: are two viruses worse than one? Med Care. 2006 Feb;44(2):158-66. doi: 10.1097/01.mlr.0000197027.06808.e2. PMID 16434915
- [Result] Jacobson CJ Jr., Luckhaupt SE, DeLaney S, Tsevat J. Religio-biography, coping, and meaning-making among persons with HIV/AIDS. Journal for the Scientific Study of Religion. 2006;45:39-56.